CLINICAL TRIAL: NCT00088868
Title: A Phase I Study Of 17-Dimethylaminoethylamino-17-demethoxygeldanamycin (17DMAG) With Evaluation Of Hsp90 Client Proteins In Subjects With Solid Tumors And Lymphomas
Brief Title: 17-Dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) in Treating Patients With an Advanced Solid Tumor or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 040218; 04-C-0218; NCI-6544; CDR0000377488; NCT00086008 (obsolete NCT alias)
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Lymphoma; Small Intestine Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; anaplastic large cell lymphoma; intraocular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult Hodgkin lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; angioimmunoblastic T-cell lymphoma; small intestine lymphoma; Waldenström macroglobulinemia; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic; Intraocular Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Mycosis Fungoides; Sezary Syndrome; Immunoblastic Lymphadenopathy; Waldenstrom Macroglobulinemia; Lymphoma, T-Cell, Cutaneous; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma

INTERVENTIONS:
Drug: alvespimycin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG), work in different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of 17-DMAG in treating patients with an advanced solid tumor or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) in patients with an advanced malignant solid tumor or lymphoma.
* Determine the dose-limiting toxic effects and toxicity profile of this drug in these patients.

Secondary

* Compare the effects of this drug on heat shock protein 90 (Hsp90) client proteins when assayed in peripheral blood mononuclear cells (PBMC) vs tumor tissue from patients treated with this drug.
* Correlate disturbances in key signaling pathways with administration of this drug in these patients.
* Determine the dose that alters key proteins in the majority of patients treated with this drug.
* Correlate serum proteomic patterns with target interactions or DMAG clinical effects in patients treated with this drug.
* Determine the pharmacokinetics of this drug in these patients.

OUTLINE: This is a single-center, dose-escalation study.

Patients receive 17-dimethylaminoethylamino-17-demethoxygeldanamycin (17-DMAG) IV over 1-2 hour on days 1 and 4 or days 2 and 5 weekly for 4 weeks. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 patients receive escalating doses of 17-DMAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of up to 6 patients experience dose-limiting toxicity. Once the MTD is determined, 10 additional patients are treated at the MTD.

PROJECTED ACCRUAL: Approximately 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant solid tumor OR lymphoma

  * Metastatic or unresectable disease
* Standard curative or palliative measures are not available OR are associated with minimal survival benefit
* No known brain metastases

  * Treated brain metastases allowed provided they have been stable ≥ 6 months without steroids or anti-seizure medications

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3
* Hemoglobin > 8 g/dL

Hepatic

* AST and ALT ≤ 2 times upper limit of normal
* Bilirubin ≤ 1.5 times normal
* PT and PTT ≤ 1.5 times normal (unless due to the presence of lupus anticoagulant or stable anticoagulation)

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No orthostatic hypotension > grade 2 (requiring more than brief fluid replacement or other therapy OR with physiological consequences)
* No New York Heart Association class III or IV heart failure
* LVEF ≥ 40% by MUGA
* QTc ≤ 450 msec (470 msec for women)
* No congenital long QT syndrome
* No myocardial infarction within the past year
* No active ischemic heart disease within the past year
* No history of uncontrolled dysrhythmias
* No history of serious ventricular arrhythmia (ventricular fibrillation or ventricular tachycardia > 3 premature ventricular contractions in a row)
* Not requiring antiarrhythmic drugs
* No poorly controlled angina
* No left bundle branch block

Pulmonary

* No uncontrolled symptomatic pulmonary disease, including any of the following:

  * Dyspnea off or on exertion
  * Paroxysmal nocturnal dyspnea
  * Severe chronic obstructive/restrictive pulmonary disease requiring daily chronic medications and oxygen
* Must not meet the Medicare criteria for home oxygen
* No sufficiently compromised pulmonary status as measured by baseline pulmonary function tests and DLCO

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation
* No known HIV positivity
* No hyponatremia indicated by sodium < 130 mmol/L
* No known immunodeficiency syndromes
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to 17-dimethylaminoethylamino-17-demethoxygeldanamycin (geldanamycin or 17-AAG)
* No concurrent uncontrolled illness
* No active or ongoing uncontrolled infection
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biologic therapy and recovered
* No concurrent prophylactic growth factors

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin, 8 weeks for UCN-01) and recovered

Endocrine therapy

* See Disease Characteristics
* Concurrent hormonal therapy for prostate cancer allowed provided patient has metastatic disease that has progressed despite prior hormonal therapy

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy that included the heart in the field (e.g., mantle radiotherapy)

Surgery

* At least 4 weeks since prior major surgery

Other

* At least 2 weeks since prior participation in a phase 0 study
* Concurrent bisphosphonates for any cancer allowed
* Concurrent preventative doses of aspirin or non-steroidal anti-inflammatory drugs allowed
* No concurrent drugs that may prolong QTc interval
* No concurrent full anticoagulation on a regular basis
* No concurrent prophylactic antiemetics
* No other concurrent investigational agents or therapies
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2004-06; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, MD, Principal Investigator — NCI - Medical Oncology Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States